CLINICAL TRIAL: NCT00370643
Title: Intensive Glucose Control Versus Conventional:Tendency Of Better Clinical Outcome In Open Heart Surgery
Brief Title: Glucose Control in Open Heart Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: number: 637-02
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Hyperglycaemia During Perioperative Period; Heart Valve Diseases; Ventricular Dysfunction
Keywords: hyperglycaemia; open heart surgery; intensive care unit
MeSH Terms: conditions — Heart Valve Diseases; Ventricular Dysfunction; Hyperglycemia | interventions — Insulin

INTERVENTIONS:
Drug: human regular insulin

SUMMARY:
The purpose of the study is to seek if there is difference to state glucose level in 80-120mg/dl or 200mg/dl in patients submitted to open heart surgery

DETAILED DESCRIPTION:
Hyperglycaemia in the intensive care unit and perioperative period has been accused to be one of the causes of worse clinical outcome. It is known that in open heart surgeries the glucose level must be set less than 200mg/dl, but new trials had set the glucose level lower than that: 140mg/dl in some studies and even lower (80-110mg/dl). Our trial had the intention to seek if there is difference setting glucose level in 2 different ones would modifies clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* adult more than 21 years old
* open heart surgery with cardiopulmonary bypass

Exclusion Criteria:

* renal dysfunction
* reoperation
* use of inotropic support
* neurological dysfunction
* chronic pulmonary obstructive disease
* emergency or urgency

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98
Dates: Start 2002-10; Study Completion 2004-11

PRIMARY OUTCOMES:
Duration of intubation
ICU length
Blood transfusion
Infection rate
Renal dysfunction
Neurological dysfunction
Hospital length
Mortality

SECONDARY OUTCOMES:
Length of surgery
Length of cardiopulmonary bypass
Physical status
EuroSCORE
Parsonnet
Canadian Multicenter index

CONTACTS AND LOCATIONS:
Overall Officials: Jose O Costa Auler Junior, Professor, Principal Investigator — Heart instutute, Hospital of Clinics, São Paulo University Medical School; Raquel PC Chan, Study Chair — Heart Institute, Hospital of Clinics, São Paulo University Medical School
Locations (1):
- Heart Institute, Hospital of Clinics, São Paulo University Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Result] Zerr KJ, Furnary AP, Grunkemeier GL, Bookin S, Kanhere V, Starr A. Glucose control lowers the risk of wound infection in diabetics after open heart operations. Ann Thorac Surg. 1997 Feb;63(2):356-61. doi: 10.1016/s0003-4975(96)01044-2. PMID 9033300
- [Derived] Chan RP, Galas FR, Hajjar LA, Bello CN, Piccioni MA, Auler JO Jr. Intensive perioperative glucose control does not improve outcomes of patients submitted to open-heart surgery: a randomized controlled trial. Clinics (Sao Paulo). 2009;64(1):51-60. doi: 10.1590/s1807-59322009000100010. PMID 19142552